CLINICAL TRIAL: NCT04494087
Title: Potential Benefit in Information Providing and Influence on Patient Anxiety and Satisfaction by Means of Preoperative Explanatory Videos in Total Extraperitoneal Inguinal Hernioplasty: a Multicenter Randomized Controlled Trial
Brief Title: The Effect of Preoperative Explanatory Videos in Total Extraperitoneal Inguinal Hernioplasty on Information Providing: a Multicenter Randomized Controlled Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 2020-01548
Record Dates: First submitted 2020-07-13; First posted 2020-07-31 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; informed consent; STAI; ICF; State-Trait Anxiety Inventory; Individual Clinician Feedback
MeSH Terms: conditions — Hernia, Inguinal | interventions — Consent Forms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Hernia video (Active Comparator): The video of the intervention group will provide a short (< 5 min) summary explaining the basic principles of endoscopic extraperitoneal hernia repair, its possible complications and the postoperative course. After carefully watching the video, participants should be able to correctly answer to a multiple-choice test consisting of 12 questions related to the aforementioned topics.
  Interventions: Other: Explanatory video
- Mock video (Placebo Comparator): This video is a general documentation of the "typical" day of surgery in the day clinic. The information is essentially limited to the pictorial representation of the individual wards which the patient will pass through during the operation (arrival at the clinic, admission, transport to the operating theatre, recovery room, discharge).
  The video explicitly does not transport any information that could be helpful for answering the quiz questions or for medical understanding of the operation itself.
  Interventions: Other: Explanatory video
- Control group (Sham Comparator): The link of the third group leads to a digital version of the information sheet, which has already been discussed with all patients during the informed consent discussion. The digital version of the informed consent form allows the patient to read the information again. The third group thus corresponds to the standard of care.
  Interventions: Other: Informed consent form

INTERVENTIONS:
Other: Explanatory video — Links to explanatory videos handed out to patients to be watched at home after standard informed consent giving
  Arms: Hernia video; Mock video
Other: Informed consent form — Links to a digital version of the informed consent form already discussed during the process of informed consent giving.
  Arms: Control group

SUMMARY:
The use of electronic media in informed consent giving has become increasingly important in recent years. Due to the easy access to information via electronical media, patients are primed in a heterogeneous manner concerning expectations and wishes regarding surgical interventions. Inherent to its nature elective interventions are critically questioned as there is time for information gathering and reflection.

In this study, the investigators set out to investigate the effect of an educational video as a supporting element in the process of informed consent giving for one the most frequently performed interventions in general surgery, namely inguinal hernia repair.

In a multi-center setup, eligible patients for primary inguinal hernia repair will be randomly assigned to 1 of 3 groups. The intervention video provides basic principles of endoscopic extraperitoneal hernia repair. The second video is similar in length and design and displays general aspects of day surgery in the two study centres. The third group's link will lead to the digital version of the informed consent. Primary outcomes will consist of 1) score in a multiple choice test assessing gain of knowledge regarding hernia repair, 2) difference in the State-Trait Anxiety Inventory (STAI) and 3) patient satisfaction questionnaire (ICF, Picker Institute, Germany) as assessed 1-2 days after the first consultation.

ELIGIBILITY:
Inclusion Criteria:

* unilateral or bilateral hernia with indication for surgical therapy
* signed informed consent form for trial participation

Exclusion Criteria:

* Patients who have had surgery for ipsi- or contralateral inguinal or femoral hernia
* combination interventions (umbilical and inguinal hernia repair, e.g.)
* cognitive, audio-visual or linguistic handicap raising concern of complete understanding of the research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 183 (Estimated)
Dates: Start 2022-05-18 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Score in multiple-choice-test | assessed 1-2 days after group allocation/exposure
  Quiz with questions regarding background, indication, implementation, complications and postoperative course of the total extraperitoneal inguinal h ernioplasty (TEP) procedure. The questions asked check relevant aspects for the patient with regard to the planned operation. The structure of the multiple-choice quiz takes the "single best option" out of 12 questions. Maximum value of the test is 12 (12/12, highest score-best outcome), the lowest 0 (0/12, lowest score-worst outcome).
  The questions are clearly posed and the correct answer is based on current guidelines for the management of inguinal hernia, which have been published by the European Hernia Society (EHS), American Hernia Society (AHS), International Endo Hernia Society (IEHS) and the European Association for Endoscopic Surgery and Other Interventional Techniques (EAES) as a consensus document by "HerniaSurge".

SECONDARY OUTCOMES:
Spielberg State-Trait Anxiety Inventory (STAI) | assessed 1-2 days after group allocation/exposure
  To test the effect of the intervention on anxiety before surgery, an anxiety score is determined using the Spielberg State-Trait Anxiety Inventory (STAI).
  The inventory is based on a 4-point Likert scale and consists of 40 questions on a self-report basis.
  Scores range from 20 to 80 with higher scores indicating greater anxiety.
Individual Clinician Feedback (ICF) | assessed 30 days postoperatively at follow-up visit
  Patient satisfaction with regard to doctor-patient communication is recorded by the validated ICF questionnaire.
  The ICF questionnaire (Picker Institute) comprises 38 items concerning the patient's experience of the examination atmosphere, the comprehensibility of the physician's statements, the participation in decisions, the course of the conversation as well as socio-demographic characteristics of the patient. The items are assessed on an 11-point Likert scale from 0 to 10, with 0 as the most critical and 10 as the most positive experience.
Numerical rating scale (NRS) | assessed 3 months postoperatively
  To assess the effect on chronic pain, the pain is assessed by telephone using the NRS score approximately 3 months after the operation.
  The numerical rating scale (NRS) requires the patient to rate his or her pain on a scale from 0 to 10, in which 0 is no pain (best outcome) and 10 the worst pain imaginable (worst outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Christian Gingert, MD, Principal Investigator — Cantonal Hospital Winterthur, Department of Surgery
Locations (2):
- Switzerland (2):
  - GZO Spital Wetzikon, Wetzikon
  - Cantonal Hospital Winterthur, Department of Surgery, Winterthur

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) with other researchers.

REFERENCES:
- [Derived] Lunger F, Frank F, Peros G, Lunger A, Vuille-Dit-Bille R, Guglielmetti L, Breitenstein S, Grieder F, Ehlers J, Gingert C. Potential benefit in information providing and influence on patient anxiety and satisfaction by means of preoperative explanatory videos in total extraperitoneal inguinal hernioplasty: study protocol of a multicentre, double-blinded, randomised parallel-group controlled trial. BMJ Open. 2021 Jan 26;11(1):e043702. doi: 10.1136/bmjopen-2020-043702. PMID 33500291